CLINICAL TRIAL: NCT03273127
Title: A Phase 1, Randomized, Single-Blind, Placebo Controlled Study to Assess Pharmacokinetics, Safety and Tolerability of Abediterol Administered Once Daily for 9 Days, in Patients With Asthma on Inhaled Corticosteroids
Brief Title: To Assess the Pharmacokinetics, Safety and Tolerability of Abediterol Administered Once Daily for 9 Days, in Patients With Asthma on Inhaled Corticosteroids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6540C00006
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Asthma, placebo, abediterol, DPI, corticosteroids
MeSH Terms: conditions — Asthma | interventions — 5-(2-((6-(2,2-difluoro-2-phenylethoxy)hexyl)amino)-1-hydroxyethyl)-8-hydroxyquinolin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is single-blind with regard to treatment (abediterol or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abediterol 5 μg (Experimental): Out of 12 randomized patients, 9 will receive abediterol 5 μg as dry inhalation powder orally once daily for 9 days. Patients will be provided salbutamol as rescue medication for use throughout the study. During the treatment period, all patients will be continued on their current ICSs. In addition, each patient will receive Abediterol 5.0 μg QD.
  Interventions: Drug: Abediterol
- Placebo (Placebo Comparator): Out of 12 randomized patients, 3 will receive placebo as dry inhalation powder orally once daily for 9 days. Patients will be provided salbutamol as rescue medication for use throughout the study. During the treatment period, all patients will be continued on their current ICSs. In addition, each patient will receive placebo QD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abediterol — A β2-adrenoceptor agonists, produce smooth muscle relaxation in the airways and improves lung function.
  Arms: Abediterol 5 μg
Drug: Placebo — Abediterol matching placebo without any pharmacological activity.
  Arms: Placebo

SUMMARY:
A Phase 1 study to assess pharmacokinetics (PK) and safety of abediterol 5 μg dry powder inhaler (DPI) given once daily (QD) for 9 days, compared to placebo, in patients with asthma on inhaled corticosteroids (ICSs).

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled study to assess PK and safety of abediterol 5 μg DPI given QD for 9 days, compared to placebo, in patients with asthma on ICSs. It is planned that 12 patients with asthma will be randomized into the study, of which 9 will receive abediterol 5 μg and 3 will receive placebo. The entire study period is scheduled to take a maximum of 41 days (follow-up included) for each individual patient. During the screening period, all patients will take their own baseline inhaled corticosteroids. Patients on long-acting β2-agonist/inhaled corticosteroids will be switched over to the respective inhaled corticosteroid mono-component at Visit 1. Patients will be provided salbutamol as rescue medication for use throughout the study. Each patient will receive a single inhaled dose of abediterol or placebo in the morning of Days 1 to 9 (Visits 3 to 8) under supervision of the Investigator or designee.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Male and non-pregnant, non-lactating female patients aged 18 - 55 years with asthma and with suitable veins for cannulation or repeated venipuncture.
* Non-smoker or former smoker who quit ≥ 6 months prior to Visit 1 and have a total smoking history of ≤ 10 pack-years. Note: Pack-years are calculated by dividing the number of cigarettes smoked per day by 20 (the number of cigarettes in a pack) and multiplying this figure by the number of years a person has been smoking. For example, a person who smokes 40 cigarettes a day and has been smoking for 10 years would have a 20 pack-year smoking history (40 cigarettes per day ÷ 20 cigarettes per pack = 2; 2 × 10 years of smoking = 20 pack-year history).
* Patient with documented clinical diagnosis of asthma for ≥ 6 months before Visit 1 according to Global Initiative for Asthma (GINA) guidelines.
* Patient with blood pressure (defined as systolic blood pressure [SBP] ≥ 90 and ≤ 140 mmHg, and diastolic blood pressure [DBP] ≥ 50 and ≤ 90 mmHg) at Screening, measured after resting in the supine position for 5 minutes.
* Patient with no relevant clinical laboratory findings at Screening (Visits 1 or 2) as judged by the Investigator.
* Patient on stable dose of ICSs for at least 1 month prior to Visit 1. Patients on bronchodilators will need to do appropriate wash-out prior to the pulmonary function test at Visit 2.
* Patient with pre-bronchodilator forced expiratory volume in 1 second (FEV1) at Visit 2 ≥ 40% and ≤ 90% of predicted (mean of 2 pre-bronchodilator measurements taken 30 minutes apart).
* Patient who demonstrates the ability to use the study inhalation device properly.

Patient able to perform acceptable pulmonary function testing for FEV1 according to American Thoracic Society (ATS)/European Respiratory Society (ERS) acceptability criteria.

* Negative pregnancy test (serum pregnancy test at Screening) for female patients.

  * Female patients must be post-menopausal, surgically sterile, or must be able to adhere to the conditions of contraceptive requirements. Male patients must be surgically sterile or must be able to adhere to the conditions of contraceptive requirements.
* Patients willing not to donate blood during the study and for 3 months following their last dose of IMP.
* Patient willing and able to follow study directions and restrictions.
* Patient must be able to read, speak and understand German language.

Exclusion Criteria:

* Patient has known or suspected hypersensitivity to the IMP or excipients, including lactose (Note: lactose intolerance is not an exclusion criterion).
* Patient who has used systemic steroid in the 6 weeks before Visit 1.
* Patient with a history of hospitalization due to asthma in the 6 months prior to Visit 1 or a history of intubation because of asthma at any time in their lifetime.
* Patient with any active pulmonary disease other than asthma.
* Patient non-compliant with study procedures in the Screening period (prior to randomization) -as judged by the Investigator.
* Patient under treatment with biologicals such as monoclonal antibodies or chimeric biomolecules including omalizumab, mepolizumab, and reslizumab within 6 months or 5 half-lives before Visit 1, whichever is longer.
* Patient treated with any investigational drug within 30 days (or 5 half-lives, whichever is longer) prior to Visit 1.
* Patient on treatment with strong cytochrome P450 (CYP)3A4 inhibitors such as ketoconazole or itraconazole or CYP3A4 inducers such as rifampin at Visit 1 or within 14 days prior to administration of IMP.
* Patient with a history, laboratory abnormality, or clinical suspicion of any clinically relevant disease or disorder, including uncontrolled hypertension or uncontrolled diabetes, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study, or any other safety concerns in the opinion of the Investigator.
* Patient with diagnosis of any kind of chronic hepatitis or known human immunodeficiency virus (HIV) infections at the time of enrolment.
* Patient with any active malignancy or treatment thereof within the five years prior to enrolment.
* Patient with any clinically important abnormalities in rhythm, conduction, or morphology of the screening 12-lead ECG as judged by the Investigator on the screening ECG.
* Patient with prolonged QT interval using Fridericia's correction ≥ 450 msec for males and females on the screening ECG or family history of long QT syndrome.
* Patient with PR (PQ) interval prolongation (> 240 msec), intermittent second or third degree atrio-ventricular (AV) block or AV dissociation or with QRS interval ≥ 120 msec or any other ECG abnormality which might affect the evaluation of the central ECG reading on the screening ECG.
* Patient with heart rate (HR) < 45 beat per minute (bpm) or > 90 bpm at Screening ECG.
* Patient with implanted cardiac defibrillator and patients with sustained symptomatic ventricular and/or atrial tachyarrhythmia.
* Patient with any contraindication against the use of sympathomimetic drugs as judged by the Investigator.
* Patient with unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society Class II, or a myocardial infarction, or stroke within 6 months before Visit 1.
* Patient with a history of hospitalization within 12 months caused by heart failure or a diagnosis of heart failure higher than New York Heart Association (NYHA) Class II.
* Patient who failed the screening procedures or patient with previous participation in the current study. Patients who failed the screening procedures may be re-screened once only.
* Patient with a history of or current alcohol or drug abuse (including marijuana), as judged by the Investigator.
* Patient with planned in-patient surgery, major dental procedure or hospitalization during the study.
* Patient involved in the planning and/or conduct of the study (applies to both AstraZeneca staff, contract research organization (CRO) staff and/or staff at the study site).
* Vulnerable person (e.g., person kept in detention).
* Patient with exacerbation requiring emergency room visit or systemic steroid use or increased dose of ICS within the Screening Period
* Patient who intends to use any concomitant medication not permitted by this protocol.
* Patient who received live attenuated vaccine within 30 days prior to Visit 1 or who received inactivated vaccine within 7 days prior to Visit 1.
* Donation or loss of > 400 mL blood and plasma within the previous 3 months prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) assessment for abediterol on Day 1 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours
  To assess Cmax after single inhaled dose of abediterol 5 μg. Cmax will be taken directly from the individual concentration-time curve.
Time to reach maximum plasma concentration (tmax) assessment for abediterol on Day 1 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours
  To assess tmax after single inhaled dose of abediterol 5 μg. tmax will be taken directly from the individual concentration-time curve.
Area under the plasma concentration-curve from time zero to the time of last quantifiable concentration (AUClast) assessment for abediterol on Day 1 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours
  To assess AUClast after single inhaled dose of abediterol 5 μg.
Area under the plasma concentration-curve from time zero to 24 hours post-dose (AUC(0-24)) assessment for abediterol on Day 1 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours
  To assess AUC(0-24) after single inhaled dose of abediterol 5 μg.
Observed maximum concentration (Cmax) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess Cmax after multiple once daily inhaled doses of abediterol 5 μg. Cmax will be taken directly from the individual concentration-time curve.
Time to reach maximum concentration (tmax) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess tmax after multiple once daily inhaled doses of abediterol 5 μg. tmax will be taken directly from the individual concentration-time curve.
Terminal rate constant, estimated by log-linear LS regression of the terminal part of the concentration-time curve (λz) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess λz after multiple once daily inhaled doses of abediterol 5 μg.
Terminal half-life, estimated as (ln2)/λz (t½λz) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess t½λz after multiple once daily inhaled doses of abediterol 5 μg.
Area under the plasma concentration-curve from time zero to the time of last quantifiable concentration (AUClast) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess AUClast after multiple once daily inhaled doses of abediterol 5 μg.
Area under the plasma concentration-curve from time zero to 24 hours post-dose (AUC(0-24)) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess AUC(0-24) after multiple once daily inhaled doses of abediterol 5 μg.
Apparent clearance for drug estimated as dose divided by AUC0-24 (CL/F) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess CL/F after multiple once daily inhaled doses of abediterol 5 μg.
Average plasma concentration during a dosing interval, estimated as AUC0-24/24 (Cavg) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess Cavg after multiple once daily inhaled doses of abediterol 5 μg.
Fluctuation index during a dosing interval estimated as 100*(Cmax - Cmin)/Cavg (%), where Cmin is the minimum concentration at the end of the dosing interval (%Fluctuation) assessment for abediterol on Day 9 | Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess %Fluctuation after multiple once daily inhaled doses of abediterol 5 μg.
Accumulation ratio for Cmax estimated as (Cmax on Day 9/Cmax on Day 1) (Rac (Cmax)) assessment for abediterol on Day 9 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours; Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess Rac (Cmax) after multiple once daily inhaled doses of abediterol 5 μg.
Accumulation ratio for AUC0-24 estimated as (AUC0-24 on Day 9/AUC0-24 on Day 1) (Rac (AUC0-24)) assessment for abediterol on Day 9 | Day 1: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12 and 24 hours; Day 9: pre-dose and post-dose at 5, 15, 30, 45 minutes and 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours
  To assess Rac (AUC0-24) after multiple once daily inhaled doses of abediterol 5 μg.
Vital sign (Blood pressure [BP]) | Change from baseline up to Day 13
  Systolic and diastolic BP (in mmHg) will be measured after the patient has rested in the supine position for at least 5 minutes and before taking any blood sample and conducting any spirometry.
Vital sign (pulse) | Change from baseline up to Day 13
  Pulse (beats per minute [bpm]) will be measured after the patient has rested in the supine position for at least 5 minutes and before taking any blood sample and conducting any spirometry.
12-lead Electrocardiograms (ECGs) including high precision QTc analysis and telemetry | Change from baseline up to Day 13
  12-Lead ECG results performed for safety evaluation will be listed for each patient and will include the ECG parameters (where applicable [Screening, pre-dose Day 1 and Follow-up]) and changes from baseline, assessment by the Investigator (normal/abnormal not clinically significant/abnormal clinically significant) and details of any abnormalities (rhythm, ectopy, conduction, morphology, myocardial infarction, ST segment, T wave and U wave observations).
Clinical laboratory assessments (hematology, clinical chemistry and urinalysis) | Change from baseline up to Day 11
  Hematology and clinical chemistry values (including serial potassium and glucose) will be listed by patient and time point including changes from baseline (pre-dose Day 1) and repeat/unscheduled measurements. Urinalysis will include glucose, protein, blood, leucocytes, flow cytometry, microscopy.
Number of patients with Adverse Events (AEs) | Change from baseline up to follow-up (14 ± 2 days post (final) dose)
  An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, electrocardiogram). In clinical studies an AE can include an undesirable medical condition occurring at any time after the patient has signed informed consent, including run-in or washout periods, even if no specific treatment has been administered.

OTHER OUTCOMES:
Exploratory Data: Change from baseline in trough forced expiratory volume in 1 second (FEV1) on Day 2 and Day 10 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose. Note: The post-dose measurements of Day 1 and Day 9 will be done on Day 2 and Day 10.
  The trough FEV1 will be defined as the mean value of the 2 measurements performed 23:15 hours and 23:45 hours after investigational medicinal product (IMP) administration on Day 1, and Day 9.
Exploratory data: Change from baseline in peak FEV1 at each time point, compared to placebo at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  The peak FEV1 will be defined as the highest measurement on Day 1, and Day 9 from the data obtained between 0 and 4 hours post-dose.
Exploratory data: Change from baseline in trough FEV1 at each time point, compared to placebo at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  The trough FEV1 will be defined as the mean value of the 2 measurements performed 23:15 hours and 23:45 hours after IMP administration on Day 1, and Day 9.
Exploratory data: Change from baseline in FEV1 AUC0-4 at each time point, compared to placebo at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  To assess FEV1 in terms of AUC (area under the curve, normalized for time) at pre-dose, at least one value between 0 and 2 hours and the value at 4 hours post-dose to calculate the normalized AUC0-4 (the area under the curve from time zero to 4 hours post-dose).
Exploratory data: Change from baseline in FEV1 AUC0-12 at each time point, compared to placebo at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  To assess FEV1 in terms of AUC at pre-dose, at least one value between 0 and 4 hours and the value at 12 hours post-dose to calculate the normalized AUC0-12 (the area under the curve from time zero to 12 hours post-dose).
Exploratory data: Change from baseline in FEV1 AUC0-24 at each time point, compared to placebo at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  To assess FEV1 in terms of AUC at pre-dose, at least one value between 0 and 12 hours and at least one value post 12 hours post-dose to calculate the normalized AUC0-24 (area under the curve from time zero to 24 hours post-dose).
Exploratory data: Time to peak FEV1 at Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  The peak FEV1 will be defined as the highest measurement on Day 1, and Day 9 from the data obtained between 0 and 4 hours post-dose.
Exploratory data: Change from baseline in FEV1 at each time point on Day 1 and Day 9 | Days 1 and 9: 45 and 15 minutes pre-dose and 15 minutes, 1, 4, 12, 23:15 and 23:45 hours post-dose.
  Change from baseline in FEV1 value at Day 1 and Day 9 will be the value difference between the calculated trough FEV1 value and the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.med. Rainard Fuhr, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany